CLINICAL TRIAL: NCT05718050
Title: Mandibular Flexure: An In-vivo Study in Dentate Patients.
Brief Title: Mandibular Flexure in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Carosi, Assistant Professor, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018065
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mandibular Flexure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexure (Experimental): Dentate patients, 18 years of age or older, in good health and, in need of implant treatment
  Interventions: Diagnostic Test: Mandibular flexure evaluation

INTERVENTIONS:
Diagnostic Test: Mandibular flexure evaluation — A mandibular silicon impression was taken, and a vacuum molded thermoplastic stent with radiopaque fiducial markers (steel ball bearings) on the facial side of the canines and molars was fabricated for each patient. Two Cone Beam Computed Tomographs (CBCTs) were made per patient with their radiographic stent in the mouth at the OVD and MO positions at the University Advanced Digital Diagnostic Center. The CBCT examination was performed without any stitching procedure using a computed tomography (SCANORA 3DX; Dexis LLC) set up at 90 kV, 4 mA and a field of view (FOV) of 140 and 100 mm in height and width respectively, to decrease the radiation dose without affecting the quality of the examination.

SUMMARY:
The flexion of the mandible (MF) is a multifactorial phenomenon that occurs simultaneously with mandibular movements determining changes in the shape of the mandible. mandibular flexure (MF) may cause complications and failures in both conventional and implant-supported fixed dental prostheses (FDP) especially when a long-span prosthesis is planned to connect the anterior to the posterior region of the mandible. Previous studies reported increased biomechanical stress at the prosthetic and implant level, poor passivity of fit, impression distortion, pain during function, de-cementation of the prosthesis, porcelain chipping, prosthetic screw loosening and fracture, bone resorption and implant fracture. The aim of this study is to quantify the dimensional changes related to MF by means of a cone beam computed tomography (CBCT) between maximum opening (MO) and maximum intercuspation (OVD) positions. The null hypothesis was that there is no significant difference in terms of length and width of the mandible between maximum intercuspation and maximum opening positions.

ELIGIBILITY:
Inclusion Criteria:

* Dentate patients,
* 18 years of age or older,
* Good health
* Need of implant treatment

Exclusion Criteria:

* active periodontitis with tooth mobility
* neuromuscular disorders
* temporomandibular joint disorders
* parafunctional habits
* systemic condition preventing surgery
* history of oro-maxillofacial radiation therapy
* history of drug or alcohol abuse
* heavy smoking
* uncontrolled diabetes
* pregnancy
* lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Mandibular Flexure in Occlusal Vertical Dimension (OVD) | 24 hours
  A blind assessor made 4 four measurements per patient on an implant planning software (DTX Studio Implant software, Dexis LLC), evaluating the distance between the fiducial landmark at the contralateral canines and contralateral molars, and between ipsilateral canines and molars on both sides
Mandibular Flexure in maximum opening (MO) | 24 hours
  A blind assessor made 4 four measurements per patient on an implant planning software (DTX Studio Implant software, Dexis LLC), evaluating the distance between the fiducial landmark at the contralateral canines and contralateral molars, and between ipsilateral canines and molars on both sides

CONTACTS AND LOCATIONS:
Locations (1):
- Benemérita Universidad Autónoma de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No